CLINICAL TRIAL: NCT07278908
Title: Efficacy and Safety of Avatrombopag Versus Avatrombopag Combined With All-trans Retinoic Acid in the Treatment of Primary Immune Thrombocytopenia: a Multicenter, Open-label, Randomized Controlled Study
Brief Title: Avatrombopag Combined With All-trans Retinoic Acid in the Treatment of Primary Immune Thrombocytopenia
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025121
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: ITP - Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia; all trans retinoic acid; Avatrombopag
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avatrombopag+All trans retinoic acid (Experimental)
  Interventions: Drug: Avatrombopag+All trans retinoic acid
- Avatrombopag (Active Comparator)
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag+All trans retinoic acid — Avatrombopag, po, starting dose 20mg qd, later adjusted dose or frequency according to response; All trans retinoic acid, po, 10mg bid.
  Arms: Avatrombopag+All trans retinoic acid
Drug: Avatrombopag — Avatrombopag, po, starting dose 20mg qd, later adjusted dose or frequency according to response
  Arms: Avatrombopag

SUMMARY:
This study is an open label, randomized controlled, multicenter clinical trial aimed at comparing the efficacy and safety of the combination of atorvastatin and all trans retinoic acid with atorvastatin alone in the treatment of first-line ineffective or recurrent immune thrombocytopenia.

The study is divided into a screening period (2 weeks), a treatment period (0-24 weeks), a reduction period (25-36 weeks), and a follow-up period (37-52 weeks), with a total of one year from the start of treatment to the end of follow-up (52 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. The patient signs an informed consent form;
2. ≥ 18 years old;
3. The patient's history of ITP is at least 3 months (persistent or chronic ITP);
4. The platelet count of the subject within 24 hours before the first administration of the study drug is less than 30 × 10^9/L; during the screening period, platelet count is measured at least twice (at least 1 week apart), with an average platelet count of less than 30 × 10^9/L and no platelet count greater than 35 × 10^9/L;
5. First line treatment, such as ineffective hormone or immunoglobulin therapy, or ITP patients who relapse after treatment;
6. Receive concomitant therapy drugs (including stable doses of glucocorticoids within the past month, stable doses of azathioprine, danazol, cyclosporine A, or mycophenolate mofetil within the past three months) for treatment; TPO receptor agonists should be discontinued at least 2 weeks before enrollment; Patients receiving anti-CD20 treatment should discontinue the medication six months prior to enrollment; Patients who underwent splenectomy were enrolled six months after the completion of the surgery;
7. Within the past year, there have been no heart diseases, including NYHA class III/IV congestive heart failure, drug-induced arrhythmias, or myocardial infarction;
8. Laboratory tests of coagulation function showed that the prothrombin time (PT/INR) and activated partial thromboplastin time (APTT) values did not exceed 20% of the normal reference range; No history of coagulation abnormalities except for ITP;
9. White blood cell count, absolute neutrophil count, and hemoglobin are within the normal range in the laboratory, with no abnormalities other than ITP, except for the following situations: a) Hemoglobin: If the anemia is clearly caused by iron deficiency anemia (excessive loss of blood related to thrombocytopenia) due to ITP, the subject's hemoglobin level below the lower limit of normal values can be selected for the study based on the researcher's judgment; c) Absolute neutrophil count ≥ 1.5 × 10^9/L can be included in the group;
10. The main organ function is good, that is, the liver and kidney function is good before treatment, AST and ALT are ≤ 1.5 times the upper limit of normal (ULN), total bilirubin is ≤ 1.5 times ULN, and serum creatinine is ≤ 1.5 times ULN;
11. The subjects adopted approved contraceptive methods. Female participants must be infertile (hysterectomy, bilateral salpingectomy, bilateral tubal ligation, or more than 1 year after menopause) or have the ability to conceive but have used study approved contraceptive methods during the entire study period until the end of the follow-up period, 2 weeks before the first dose; Women with fertility must have a negative serum pregnancy test within 24 hours prior to the first dose of medication;
12. The subjects fully understand and are able to comply with the requirements of the research protocol, and are willing to complete the study as planned.

Exclusion Criteria:

1. Individuals who are allergic to known ingredients or excipients in atorvastatin or all trans retinoic acid;
2. Accept medication maintenance therapy (including but not limited to aspirin, clopidogrel, and/or nonsteroidal anti-inflammatory drugs NSAIDs) or anticoagulants that affect platelet function or quantity;
3. Accompanied by autoimmune hemolytic anemia, or various secondary or hereditary thrombocytopenia; Such as leukemia, lymphoma, multiple myeloma, aplastic anemia, myelodysplastic syndrome, Evans syndrome, common variant immunodeficiency, systemic lupus erythematosus, cirrhosis, antiphospholipid antibody syndrome, pseudothrombocytopenia, drug-induced thrombocytopenia (such as quinine, heparin, antimicrobial drugs, antiepileptic drugs, etc.), etc;
4. There is bone marrow fibrosis with MF ≥ 2;
5. Participate in other research drug studies (including vaccine studies) or be exposed to other research drugs (TPO receptor agonists or salvage treatments) within 4 weeks or 5 half lives (whichever is longer) before the first use of the medication;
6. Previous ITP treatments, including rescue therapy with platelet transfusions, glucocorticoids, immunoglobulins, immunomodulators, etc., did not end within 2 weeks prior to enrollment;
7. The subject has a history of any arterial/venous thrombosis (including stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, or pulmonary embolism) within the past year;
8. Pregnant or lactating women;
9. History of alcohol/drug abuse within 12 months prior to screening or first dose;
10. Previous studies have shown poor efficacy in the treatment of sufficient and sufficient doses of atorvastatin;
11. Previous all trans retinoic acid had poor efficacy;
12. All laboratory or clinical evidence of HIV infection and active hepatitis during screening. Laboratory tests during the screening period indicate active hepatitis C infection or hepatitis B infection. (hepatitis B reference: HBsAg positive and HBV DNA ≥ 500 IU/ml; Hepatitis C reference: HCV antibody positive and HCV virus copy number>upper limit of normal);
13. Life threatening bleeding (WHO bleeding score 3) or estimated need for salvage treatment before the first dose of treatment in patients;
14. History of malignant tumors or accompanying malignant tumors;
15. The researchers believe that there are any other circumstances that may prevent the subjects from completing the study or pose significant risks to them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Free Rate at week 52 | up to 52 weeks

SECONDARY OUTCOMES:
At weeks 12 and 24 without rescue treatment, the proportion of subjects with platelet levels reaching CR, R, and ≥ 50 × 10^9/L, respectively | up to 12 and 24 weeks
Treatment Free Rate at week 12 after discontinuation of treatment | up to 12 weeks after discontinuation of treatment
The proportion of subjects whose platelet levels reached CR and R at 12 weeks after discontinuation of treatment | up to 12 weeks after discontinuation of treatment
The time from the start of treatment to the first platelet count ≥ 50 × 10^9/L | up to 52 weeks
  From date of randomization until the date of first documented platelet count ≥ 50 × 10^9/L, assessed up to 52 weeks
The time required from the start of treatment to the first platelet count increasing by at least 2 times compared to the baseline platelet count | up to 52 weeks
  From date of randomization until the date of first documented platelet count increasing by at least 2 times compared to the baseline platelet count, assessed up to 52 weeks
The number of times subjects received rescue therapy during treatment and follow-up, and the proportion of subjects who received at least one rescue therapy | up to 52 weeks
World Health Organization(WHO) bleeding scoring criteria | up to 52 weeks
  score range: 0-4; higher scores mean a worse outcome
The Functional Assessment ot Chronic Illness Therapy-Fatigure(FACITF) score | up to 52 weeks
  score range: 0-52; higher scores mean a worse outcome
Adverse event | up to 52 weeks

IPD SHARING:
Plan to Share IPD: No